CLINICAL TRIAL: NCT02764359
Title: Single-Center Prospective Study of Obese Patients Comparing Two Vancomycin Loading Dose Regimens
Brief Title: Study of Obese Patients Comparing Two Vancomycin Loading Dose Regimens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, William Payne, Emergency Medicine Physician, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-120
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Infection; Sepsis; Obesity
MeSH Terms: conditions — Infections; Sepsis; Obesity | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Vancomycin loading dose- higher (Experimental): IV Vancomycin loading dose: 20 mg/kg with a maximum dose of 4,000mg
  Interventions: Drug: IV vancomycin
- IV Vancomycin loading dose- lower (Experimental): IV Vancomycin loading dose: 20 mg/kg with a maximum dose of 2,000mg
  Interventions: Drug: IV vancomycin

INTERVENTIONS:
Drug: IV vancomycin — IV vancomycin for the treatment of infection. Following the vancomycin loading dose, vancomycin dosing will be at the discretion of the pharmacist and attending physician and will follow standard of care.

SUMMARY:
Obesity alters the movement through the body of several antibiotics, including vancomycin. Based on literature to date, total body weight should be used to determine dosages and shorter dosing intervals may be needed. However, hospitals have different approaches to managing vancomycin in this patient population. The most common example is not exceeding a dose of 2,000mg of vancomycin at one time in these patients. However, some institutions including the Charleston Area Medical Center do not have a set maximum one time dose. To date, a study has not been done comparing two different dosing regimens in obese patients to determine if having a maximum dose cap is beneficial.

This research study is attempting to add to the limited existing body of literature regarding vancomycin dosing in obese patients. The investigators hypothesize that optimizing the initial or loading vancomycin dose that obese patients receive will decrease the time to target concentrations. For this study, obese adult patients will be randomized to receive either 1) a loading dose of 20 mg/kg with a maximum dose up to 2,000mg OR 2) a loading dose of 20 mg/kg with a maximum dose of up to 4,000mg. The study's primary aim is to determine differences in the time needed to achieve target vancomycin concentrations and the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age who present to the Charleston Area Medical Center-Memorial Hospital Emergency Department
* Weight >100kg
* Infection requiring intravenous vancomycin and admission to Charleston Area Medical Center-Memorial Hospital

Exclusion Criteria:

* Any patient <18 years of age
* Patients on dialysis or with unstable renal function (a change of >0.5 mg/dL in SCr concentration in patients with a SCr of <2 mg/dL or a 20% change in SCr in patients with a SCr of ≥2 mg/dL)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-01-22 (Estimated); Study Completion 2021-01-22 (Estimated)

PRIMARY OUTCOMES:
Time to attain therapeutic vancomycin concentrations | < 7 days

SECONDARY OUTCOMES:
Reported adverse events | 48 hours post initial vancomycin dose
  Red Man's syndrome: pruritus and erythematous rash involving the face, neck, and upper torso.
  Nephrotoxicity: increase in serum creatinine (SCr) by 0.5 mg/dL or 50% from baseline on two consecutive measurements.
Examine the pharmacokinetic parameter of elimination rate constant (ke) following the loading vancomycin dose | 12 hours
Examine the pharmacokinetic parameter of volume of distribution (Vd) following the loading vancomycin dose | 12 hours
Intensive care unit length of stay | 30 days
Hospital length of stay | 30 days
In-hospital mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CAMC Health Systems, Charleston, West Virginia, United States